CLINICAL TRIAL: NCT00076739
Title: Examining Associative Relations in Structured Event Complexes Using Functional Neuroimaging
Brief Title: Study of Brain Function During Cognitive Tasks
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040113; 04-N-0113
Record Dates: First submitted 2004-02-02; First posted 2004-02-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-12

CONDITIONS: Healthy
Keywords: Prefrontal Cortex; Semantic Memory; Semantic Relations; Priming Paradigm; fMRI; Healthy Volunteer; HV

SUMMARY:
This study will use magnetic resonance imaging (MRI) to examine which areas of the brain are involved in performing certain cognitive tasks. MRI uses a strong magnetic field and radio waves to produce images of body tissues and organs that provide information about structure and function of tissues.

Healthy normal volunteers between 21 and 40 years of age may be eligible for this study. Candidates must be native English speakers and must be right-handed. They must have no history of nervous system disease or psychiatric disorder. Candidates are screened with questionnaires and a neurological examination.

Participants undergo functional MRI scanning. For this procedure, the subject lies on a stretcher that moves into the scanner - a metal cylinder surrounded by a strong magnetic field. During the scan, he or she is asked to make various decisions about whether words are related or not. Two words are presented visually, separated by a variable time delay. The subject reads both words, decides as quickly and accurately as possible whether the two words are related or not, and indicates the answer by pressing a button. The test takes about 2 hours. When it is completed, the subject completes a written questionnaire concerning his or her experience in the scanner.

...

DETAILED DESCRIPTION:
Objective. The purpose of the protocol is to extend the structured event complex (SEC) model developed by the principal investigator. Grafman (Grafman, 1995) proposed that action sequences are represented in form of SECs in the human prefrontal cortex (PFC). An SEC is a goal-oriented set of events that is sequentially structured and represents thematic knowledge, morals, abstractions, concepts, social rules, event features, event boundaries, and grammars. There are both temporal and semantic associative relations between subcomponents of SEC knowledge. We will investigate hypotheses regarding the role of different regions within the PFC in processing associative relations. We will also investigate how SECs differing in psychological dimensions such as temporal duration, complexity, and familiarity are represented and activated in the PFC. We will further examine the temporal and semantic organization of SEC subcomponents by investigating how the goal and outcome structure of event knowledge is represented and activated in the PFC. Further, we will investigate how the temporal location of events within SECs are represented and activated in the PFC. We will also investigate how goals and outcomes specifying the temporal order and duration of SEC subcomponents are processed within the PFC. Additional objectives are to (1) investigate the neural representation of human emotions and decision-making based on utility estimation; (2) investigate the relationships between cognitive and neural substrates of moral emotions and judgment (Moll et al., 2002a; Moll et al., 2002b) with those of the SEC model developed by the principal investigator (Grafman, 1995); and (3) probe a new construct of cognitive dimensions incorporating critical explanatory variables in social cognition such as moral emotions and social event knowledge.

Study Population. In nineteen separate studies, healthy, normal adult volunteers will participate in experiments dealing with different kinds of associative relations in SECs using functional magnetic resonance imaging (fMRI).

Design. The experiments we are conducting will employ within-subject, rapid event-related fMRI designs to determine whether different types of SEC associative and other types of relations are stored in dissociable networks in the PFC. In nineteen experiments; we hope to automatically activate lexical, event-based and temporally-based associative and other types of relations in SECs.

Outcome Measures. The data collected will consist of accuracy and response time measures of cognitive performance reflecting automatic priming of associative relations and fMRI activation images corresponding to each kind of associative relation, and accuracy and response time measures of cognitive performance reflecting how temporal duration, complexity, and familiarity are represented and activated. Experiments 10 and 11 will also record donation choices made by the subjects. The results gained from this protocol will provide further evidence for modifying, supporting, or rejecting aspects of the SEC model, and will provide further evidence for modifying, supporting, or rejecting aspects of a framework of social cognition such as moral behavior and social event knowledge.

ELIGIBILITY:
* INCLUSION CRITERIA:

In all the studies, subjects will consist of healthy, native English-speaking, right-handed volunteers, as measured by the Edinburgh Handedness Inventory.

Subjects will range in age from 21 to 40 years old and they will be included regardless of race or gender.

EXCLUSION CRITERIA:

Non-native English speakers and non-right handers will be excluded as mentioned above, as will non-neurologically normal volunteers.

Subjects younger than 21 and older than 40 will be excluded.

A pregnancy test will be employed with all women of childbearing age. The results must be negative in order to proceed with the MRI.

Subjects with any of the following: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body, e.g. metal shavings; permanent eyeliner; insulin pump; or irremovable body piercing will be excluded from the study due to the possible dangerous effects of the magnet upon metal objects in the body.

Subjects taking central nervous system active medications will be excluded.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 452 (Actual)
Dates: Start 2004-02-02; Study Completion 2011-12-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abernethy M, Coney J. Semantic category priming in the left cerebral hemisphere. Neuropsychologia. 1996 May;34(5):339-50. doi: 10.1016/0028-3932(95)00144-1. PMID 9148190
- [Background] Belliveau JW, Kennedy DN Jr, McKinstry RC, Buchbinder BR, Weisskoff RM, Cohen MS, Vevea JM, Brady TJ, Rosen BR. Functional mapping of the human visual cortex by magnetic resonance imaging. Science. 1991 Nov 1;254(5032):716-9. doi: 10.1126/science.1948051.
- [Background] Belliveau JW, Rosen BR, Kantor HL, Rzedzian RR, Kennedy DN, McKinstry RC, Vevea JM, Cohen MS, Pykett IL, Brady TJ. Functional cerebral imaging by susceptibility-contrast NMR. Magn Reson Med. 1990 Jun;14(3):538-46. doi: 10.1002/mrm.1910140311. PMID 2355835